CLINICAL TRIAL: NCT05885061
Title: Effects of Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UAarhus_SCS
Record Dates: First submitted 2023-05-01; First posted 2023-06-01 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Suggestion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Spinal cord stimulation turned on (Active Comparator)
  Interventions: Device: Spinal cord stimulation turned on (suggestions: off)
- Spinal cord stimulation turned off (Placebo Comparator)
  Interventions: Device: Spinal cord stimulation turned off (suggestions: on)
- Spinal cord stimulation turned on and suggestions (Active Comparator)
  Interventions: Device: Spinal cord stimulation turned on with suggestions (suggestions on)
- Control (No Intervention)

INTERVENTIONS:
Device: Spinal cord stimulation turned on (suggestions: off) — Spinal cord stimulation turned on with verbal suggestions of treatment off
  Arms: Spinal cord stimulation turned on
Device: Spinal cord stimulation turned off (suggestions: on) — Spinal cord stimulation turned off with verbal suggestions of treatment on
  Arms: Spinal cord stimulation turned off
Device: Spinal cord stimulation turned on with suggestions (suggestions on) — Spinal cord stimulation turned on with verbal suggestions of treatment on
  Arms: Spinal cord stimulation turned on and suggestions

SUMMARY:
The goal of this interventional study is to test effects of spinal cord stimulation in patients receiving treatment for their chronic pain. The main question of the study is:

• What is the effect of spinal cord stimulation when compared to placebo? Participants will rate their pain with their usual spinal cord stimulation on and off.

ELIGIBILITY:
Inclusion Criteria:

* Patients (>18 years of age) with SCS implanted to treat chronic pain.
* Patients who consent to participation and can cooperate in the study.
* Use of continuous paresthesia-free SCS for minimum 6 months prior to participation in the study.
* Pain score of 7 or less on a 0-10 scale in the most painful area treated with SCS, rated upon inclusion.
* Patients not receiving other neuromodulation treatment.
* Patients who have not undergone changes in their (pain relevant) medication during the last 30 days (pro necessitate medication allowed).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity, Visual Analogue Scale | Every 30 minutes during study session (max 5 hours)
  0-10 (0=no pain, 10=worst imaginable pain). Continual assessments to register changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No